

## **Statistical Analysis Plan (SAP)**

# Effects of low-intensity blood-flow restricted exercise compared to standard rehabilitation in patients with knee osteoarthritis

# **Trial registration**

ClinicalTrials.gov trial registration identifier:

Ethical Committee in Region Hovedstaden: H-19079135

Data Protection Agency: P-2019-814

# Statistical Analysis Plan Version and Date

Version: 1.0

Date: 30.05.2022

# **Statistical Analysis Plan Authors**

Brian Sørensen

Finn Johannsen

Per Aagaard

Peter Magnusson

Christian Couppé

Charlotte Suetta



# Signatures

| Brian Sørensen, MSc., PhD | stud. | |
|---|---|---|
| Institute of Sports Medicine | | |
| Bispebjerg Hospital | Signature: Brian Sprensen | Date: 30.05.2022 |
| Finn Elkjær Johannsen, Chie | f Physician, MD | |
| Institute of Sports Medicine | A | |
| Bispebjerg Hospital | Signature | Date: 31,05,2022 |
| Per Aagaard, Professor | | |
| Department of Sports Science | e and Clinical Biomechanics | |
| University of Southern Denn | nark | |
| | Signature: Per Alfanel | Date: 30.05.2022 |
| Peter Magnusson, Professor, | Dr.med | |
| Institute of Sports Medicine | 2 20 E 1 E | |
| Bispebjerg Hospital | Signature: 5 Peter Magur | Date:_30-05.2022 |
| Christian Couppé, PhD | | |
| Institute of Sports Medicine | | |
| Bispebjerg Hospital | Signature: Cha Couper | Date: 07-06-2022 |
| Charlotte Suetta, Professor | | |
| Department of Clinical Medi | | |
| Bispebjerg Hospital | Signature: Charlotte Suetta | 30.05.2022<br>Date: |



# **Table of Contents**

| 1. | Int | roduction | 4 |
|----|------|-----------------------------------|----|
| 1. | Stu | tudy objectivetudy objective | |
| 2. | | udy design6 | |
| | 2.1. | Intervention procedures | 6 |
| | 2.2. | Sample size calculation | 7 |
| | 2.3. | Blinding and randomization | 7 |
| 3. | Ou | itcomes | 7 |
| | 3.1. | Primary outcome | 7 |
| | 3.2. | Secondary outcomes | 8 |
| 4. | Inc | clusion and exclusion criteria | 8 |
| 5. | An | alysis | 10 |
| | 5.1. | Primary analysis | 10 |
| | 5.2. | Secondary analyses | 10 |
| | 5.3. | Intension-to-treat (ITT) analysis | 10 |
| | 5.4. | Per protocol (PP) analysis | 10 |
| 6. | Re | ferences | 11 |



30.05.2022

#### 1. Introduction

Osteoarthritis (OA) is second most common disease in Denmark and it is estimated that over 1 million Danish people suffer from OA in one or multiple joints<sup>1,2</sup>. A significant part of these people receive treatment to reduce the pain and improve the ability to work, and the socioeconomic costs in Denmark as a direct consequence of OA is estimated to be approximately 11 billion Danish kroner (1,5 million EUR) per year<sup>2</sup>.

Knee-OA is the most common OA-diagnosis and it is estimated that 60.000 Danish people with symptoms of knee-OA seek medical treatment each year<sup>3</sup>. The occurrence of knee-OA is related to overweight, inactivity, aging, earlier knee injuries, muscle weakness and exposure to lifelong physical work<sup>4-6</sup>. The elderly population continuous to increase, and so does the numbers of inactive and overweight people and therefore the occurrence of knee-OA can be expected to increase in the coming decades.

Representing the most widespread non-medical and non-operative treatment modality both internationally and in Denmark, knee-OA patients often are offered a combination of patient education, weight loss counseling and physical exercise program<sup>3,7</sup>. Physical exercise including conventional strength training, functional training (whole body exercises) and cardiovascular training all seem to have improving effects on knee pain, functional function and quality of life, respectively, in people with OA<sup>8-13</sup>. In Denmark, the GLA:D (Good Life with osteoArthritis in Denmark) concept is a nationwide exercise paradigm, which consists of eight weeks of designated and supervised multi-component training performed twice weekly<sup>14-16</sup>. The concept is a combination of education and supervised neuromuscular exercise (NEMEX) delivered by GLA:D-certified physiotherapists, with the purpose to improve lower limb muscle strength and increase muscular stability around the knee- and hip joints, respectively<sup>14-16</sup>. NEMEX has previously shown positive results on pain perception<sup>11,15-20</sup>, functional capacity<sup>11,15</sup> and quality of life<sup>15,16</sup>, however the effect of NEMEX (or GLA:D) on muscle strength and lower limb muscle mass has never been investigated to the best of our knowledge. Notably, deficits in maximal muscle strength often is often a critical factor in people with knee-OA, and can reach of 20-40 % compared to healthy sex and age-matched individuals<sup>21-23</sup>. Furthermore, prior systematic reviews have indicated that reduced knee extensor muscle strength is an important risk factor for the incidence of KOA as well as for the severity of symptoms and the decline in functional performance<sup>6,24</sup>. As such, improving lower limb muscle strength, with a particular focus on knee extensor strength,



may be a key factor in improving symptoms and function in KOA. People with OA, who are able to tolerate heavy strength training, typically experience a positive effect on maximal muscle strength and power<sup>25,26</sup>. Unfortunately however, a large proportion of OA patients are forced to refrain from this type of training due to excessive joint- and muscle pain during and following the training sessions<sup>27</sup>.

In recent years strength training combined with concurrent blood flow restriction, i.e. occlusion training, has gained increasing acceptance and usage in athletes<sup>28,29</sup> as well as different patient groups<sup>30-38</sup>. This type of training, often referred as BFR (Blood Flow Restricted) exercise, imposes low levels of mechanical load on the involved muscles and joints because the exercises are performed using low exercise loads ( $\leq 30\%$  of max) concurrently with a reduced blood flow to the working muscles, which is achieved by means of a pneumatic blood pressure cuff. BFR training has been documented to result in significant improvements in muscle mass and muscle strength even with just a few weeks of intense daily training<sup>39-41</sup>. Moreover, especially in the clinical setting, BFR exercise has been reported to effectively activate muscular satellite cells (stem cells), which are involved in muscle regeneration and myofiber growth 40,42. The marked improvements in muscle mass and strength with BFR training seem to be comparable to that achieved by conventional heavy-resistance strength training<sup>30,32,35,36,39,43</sup>. Importantly, recent data indicate that BFR can have an acute pain-reducing effect<sup>34,36</sup> and result in greater strength gains and more pronounced reductions in pain with daily activities compared to heavy strength training in knee patients who experiences pain during training<sup>31</sup>. Based on these observations BFR exercise may represent an attractive alternative training modality in patients with knee-OA.

## 1. Study objective

To investigate whether an enhanced rehabilitating effect on muscle function and joint pain can be achieved by training with low-intensity BFR exercise compared to standard rehabilitation (education and exercise) in people with knee-OA.

We hypothesise that 12 weeks of BFR training will lead to improved perceived joint pain and muscle function compared to GLA:D training.



# 2. Study design

Inclusion takes place via the Institute of Sportsmedicine (ISMC), and the Department of Physical and Occupational Therapy at Bispebjerg Hospital. Assessment for inclusion is made after referral from general practitioner or after conversation with physician assessor at the ISMC. Recruitment will also include advertising through local newspapers, posters in public libraries, social media etc., as well as invitations to attend lectures with information about the study.

Participants will be invited to a preparatory examination by the attending rheumatology chief physician at Bispebjerg Hospital. At the consultation a standard clinical assessment will be performed and the participant will be examined for meeting the explicit inclusion or exclusion criteria of the study. For participants adhering to the inclusion criteria, an information document will be handed out and the participant will be invited into an in-depth interview about the study with the chief physician. If the participant after receiving all oral and written information wishes to participate in the study and also meets the objective X-ray criteria for OA, an informed consent will be obtained. Randomization procedures will take place following baseline testing, which will be performed at Bispebjerg Hospital by a blinded (to group allocation) assessor. Subsequently, training intervention procedures will be initiated.

#### 2.1. Intervention procedures

All included patients will be randomized into two intervention groups, either standard rehabilitation (education and exercise) or BFR strength training. Each participant randomized to the education and exercise programme will be offered participation in the GLA:D programme<sup>16</sup>. GLA:D training will involve a circuit training program with four stations. Each station involves two to six exercises where the participants perform 10-15 repetitions over 2-3 sets, which depends on the participants pain- and functional level. The BFR group will perform unilateral training with the knee-OA diagnosed leg only. BFR training is performed with the BFR cuff placed at the top of the thigh on the leg being trained. The cuff will be inflated to 60-80 % of the total arterial occlusion pressure (AOP)<sup>44-48</sup>. The participant will afterwards perform training of the knee extensors in a leg press exercise machine and a leg extension exercise machine with a load corresponding to 30 % of the maximal load (1RM = Repetition Maximum)<sup>45,46,48</sup>.



The intervention period will last 12 consecutive weeks with 2 weekly training sessions at selected physiotherapy clinics. The participants in the GLA:D group will attend a supervised group training with certified GLA:D instructors. Training in the BFR group will be conducted at Bispebjerg Hospital by trained supervisors (PT) who are experienced in BFR exercise intervention. Both intervention groups will attend a 2-hours GLA:D-lecture performed by the involved physiotherapists within the first 8 weeks of training. The lecture includes information about osteoarthritis, how to deal with the diagnosis, and presenting information about ergonomics, treatment and training related to OA<sup>16</sup>.

#### 2.2. Sample size calculation

The estimated number of participants in the study are based on the primary outcome variable, KOOS-Pain subscale<sup>49</sup>, with the assumption that a change of 10 KOOS points may be considered of clinical relevance<sup>49,50</sup> as well as assuming a standard deviation (SD) averaging 15 KOOS points<sup>11,50</sup>. Assuming a statistical power of 80 %, a significance level of 0.05 and an expected within-group change in KOOS of 10 points magnitude with 12 weeks training (primary endpoint), was calculated to require 37 participants. To compensate for potential dropouts, a total of 90 participants are planned to be included in the study, divided equally and randomly into two intervention groups (45 participants in each group).

# 2.3. Blinding and randomization

The physician assessor conducting the pre and post testing of physical function, muscle mechanical function, ultrasonography and all statistical analysis will be blinded to participants' group allocation. The participants and the physiotherapists conducting both GLA:D- and BFR-training cannot be blinded for group allocation.

After baseline assessment, patients will be randomized (1:1) to either the GLA:D-training group or the BFR-training group using the Research Electronic Data Capture (REDCap) randomisation system.

#### 3. Outcomes

#### 3.1. Primary outcome

Primary outcome variable is KOOS (Knee injury and Osteoarthritis Outcome Score)
Pain subscale. KOOS is an instrument to assess the patient's opinion about their knee



and associated problems. KOOS consists of 5 subscales; Pain, Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related quality of life (QOL).

# 3.2. Secondary outcomes

Secondary outcome variables at functional level includes:

- 4x10 m maximal horizontal fast-paced walking<sup>51,52</sup>
- 30-s chair-stand test<sup>51-54</sup>
- Stair Climb test (12 steps)<sup>51,55-58</sup>
- Pain Pressure Threshold on affected and non-affected side<sup>59-64</sup>
- Total KOOS score<sup>49,50</sup>
- Oxford Knee Score<sup>49,65</sup>

Secondary outcome parameters related to mechanical muscle function will be obtained as well, including:

- Maximal isometric knee extensor (KE) strength (KinCom, isokinetic dynamometer)<sup>66-68</sup>
- KE Rapid force capacity (Rate of Force Development, RFD) (KinCom, isokinetic dynamometer)<sup>66,68,69</sup>
- Maximal leg muscle power (Nottingham Power Rig)<sup>11,69-71</sup>
- Lower limb muscle mass (Ultrasonography)<sup>72-79</sup>
- Muscle biopsies will be obtained from the thigh muscle (vastus lateralis) for evaluation of myocellular properties (myofiber area, vascularization, muscular satellite cells, myonuclei content)<sup>40,80-84</sup>

Testing will take place before the intervention period, after 8 weeks of training and at the end of the intervention (12 weeks) except for the muscle biopsies which will be obtained before the intervention period and at 12 weeks (primary endpoint). Moreover, patient-reported questionnaires and functional performance will be assessed 6 months after the intervention period.

#### 4. Inclusion and exclusion criteria

All people with symptoms of knee-OA or patients diagnosed with knee-OA are eligible. To be included in the study, participants must meet the following inclusion criteria:



- All participants must meet the American College of Rheumatology (ACR) criteria for OA<sup>85</sup>
- Visible OA on X-ray pictures (Kellgren & Lawrence grade 2-3)<sup>86</sup>
- Pain and functional limited for a minimum of 3 months
- Be able to voluntarily (i.e. unassisted) perform a 90 degrees flexion in the knee while standing
- Be able to perform loaded machine exercise (knee extension) planned for the BFR training
- Be able to understand written and spoken danish
- Be able to complete the intervention period without extensive time away

Individuals will be excluded if meeting these exclusion criteria:

- Kellgren & Lawrence grade 1 and 4<sup>86</sup>
- Bilateral OA-symptoms
- Prior knee- or hip alloplasty
- Glucocorticosteroid injection in the knee within the last 6 months
- Inflammatory arthritis
- Known neurotic disease such as multiple sclerosis or peripheral neuropathy
- Prior myocardial infarct or apoplexy, or chest pain during physical activity
- Other health related or medical conditions which makes it challenging to participate in the study

Furthermore, it is an exclusion criterium in the following conditions where use of pneumatic occlusion would be considered contraindicated:

- Type I Diabetes
- Peripheral vascular disease
- Excessive varicose veins
- Prior history of deep venous thrombosis
- Venous insufficiens causing edema in the lower legs
- Systolic blood pressure exceeding 160 mmHg or below 100 mmHg



# 5. Analysis

All outcome variables will be presented using descriptive statistics such as numerical mean and standard deviation (SD) with 95% confidence interval. Binary and categorical variables will be presented using counts and percentages. SPSS will be used for all statistical analysis. Statistician will be blinded to group allocation.

The subsections below will describe the specific procedures of statistical analyses and related descriptive statistics.

#### 5.1. Primary analysis

The change in the primary outcome (KOOS-Pain) from baseline to primary endpoint (12 weeks) will be calculated for both groups, and a mixed linear model will be used to examine if there is a systematic difference between the two intervention groups.

## 5.2. Secondary analyses

For all secondary outcomes, including the primary outcome, assessed at multiple time points (more than two) will be analysed using a mixed linear model approach. Secondary outcomes assessed at baseline and at one more time point will be analysed as described for the primary outcome above.

Explorative analysis will be conducted. The primary outcome will be correlated to the various secondary outcomes.

#### 5.3. Intension-to-treat (ITT) analysis

Statistical ITT analysis will include all subjects who are randomized to the intervention procedures.

#### 5.4. Per protocol (PP) analysis

Statistical PP analysis will include subjects who adhere to the major criteria in the protocol and completed the whole study period (i.e. all subjects with  $\geq$ 85 % training adherence).



#### 6. References

- 1. Jensen H, Davidsen M, Ekholm O, Christensen A. Danskernes Sundhed Den Nationale Sundhedsprofil 2021. *Sundhedsstyrelsen*. 2022;
- 2. Johnsen N, Kock M, Davidsen M, Juel K. De samfundsmæssige omkostninger ved artrose. *Statens Institut for Folkesundhed*. 2014;
- 3. Sundhedsstyrelsen. Knæartrose Nationale kliniske retningslinjer og faglige visitationsretningslinjer. 2012;
- 4. Ashkavand Z, Malekinejad H, Vishwanath BS. The pathophysiology of osteoarthritis. *Journal of Pharmacy Research*. 2013/01/01/2013;7(1):132-138. doi:https://doi.org/10.1016/j.jopr.2013.01.008
- 5. Silverwood V, Blagojevic-Bucknall M, Jinks C, Jordan JL, Protheroe J, Jordan KP. Current evidence on risk factors for knee osteoarthritis in older adults: a systematic review and meta-analysis. *Osteoarthritis and cartilage*. Apr 2015;23(4):507-15. doi:10.1016/j.joca.2014.11.019
- 6. Øiestad BE, Juhl CB, Eitzen I, Thorlund JB. Knee extensor muscle weakness is a risk factor for development of knee osteoarthritis. A systematic review and meta-analysis.

  Osteoarthritis and cartilage. 2015;23(2):171-177. doi:10.1016/j.joca.2014.10.008
- 7. McAlindon TE, Bannuru RR, Sullivan MC, et al. OARSI guidelines for the non-surgical management of knee osteoarthritis. *Osteoarthritis and cartilage*. Mar 2014;22(3):363-88. doi:10.1016/j.joca.2014.01.003
- 8. Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualized goal-based NEMEX-TJR training program. *BMC musculoskeletal disorders*. Jun 17 2010;11:126. doi:10.1186/1471-2474-11-126
- 9. Dantas LO, Salvini TF, McAlindon TE. Knee osteoarthritis: key treatments and implications for physical therapy. *Braz J Phys Ther*. Mar-Apr 2021;25(2):135-146. doi:10.1016/j.bjpt.2020.08.004
- 10. Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: A Cochrane Systematic Review. *Br J Sports Med.* Jan 9 2015;1:1554-7. doi:10.1002/14651858.CD004376.pub3
- 11. Holm PM, Schrøder HM, Wernbom M, Skou ST. Low-dose strength training in addition to neuromuscular exercise and education in patients with knee osteoarthritis in



secondary care - a randomized controlled trial. *Osteoarthritis and cartilage*. Jun 2020;28(6):744-754. doi:10.1016/j.joca.2020.02.839

- 12. Skou ST, Rasmussen S, Laursen MB, et al. The efficacy of 12 weeks non-surgical treatment for patients not eligible for total knee replacement: a randomized controlled trial with 1-year follow-up. *Osteoarthr Cartil*. Sep 2015;23(9):1465-75. doi:10.1016/j.joca.2015.04.021
- 13. Villadsen A, Overgaard S, Holsgaard-Larsen A, Christensen R, Roos EM. Immediate efficacy of neuromuscular exercise in patients with severe osteoarthritis of the hip or knee: a secondary analysis from a randomized controlled trial. *The Journal of rheumatology*. Jul 2014;41(7):1385-94. doi:10.3899/jrheum.130642
- 14. Roos EM, Grønne DT, Skou ST, et al. Immediate outcomes following the GLA:D® program in Denmark, Canada and Australia. A longitudinal analysis including 28,370 patients with symptomatic knee or hip osteoarthritis. *Osteoarthr Cartil*. Apr 2021;29(4):502-506. doi:10.1016/j.joca.2020.12.024
- 15. Skou ST, Odgaard A, Rasmussen JO, Roos EM. Group education and exercise is feasible in knee and hip osteoarthritis. *Danish medical journal*. Dec 2012;59(12):A4554.
- 16. Skou ST, Roos EM. Good Life with osteoArthritis in Denmark (GLA:D™): evidence-based education and supervised neuromuscular exercise delivered by certified physiotherapists nationwide. *BMC musculoskeletal disorders*. Feb 7 2017;18(1):72. doi:10.1186/s12891-017-1439-y
- 17. Bandak E, Christensen R, Overgaard A, et al. Exercise and education versus saline injections for knee osteoarthritis: a randomised controlled equivalence trial. *Ann Rheum Dis*. Nov 29 2021;doi:10.1136/annrheumdis-2021-221129
- 18. Davis AM, Kennedy D, Wong R, et al. Cross-cultural adaptation and implementation of Good Life with osteoarthritis in Denmark (GLA:D<sup>TM</sup>): group education and exercise for hip and knee osteoarthritis is feasible in Canada. *Osteoarthritis and cartilage*. Feb 2018;26(2):211-219. doi:10.1016/j.joca.2017.11.005
- 19. Holm PM, Petersen KK, Wernbom M, Schrøder HM, Arendt-Nielsen L, Skou ST. Strength training in addition to neuromuscular exercise and education in individuals with knee osteoarthritis-the effects on pain and sensitization. *Eur J Pain*. Oct 2021;25(9):1898-1911. doi:10.1002/ejp.1796
- 20. Skou ST, Bricca A, Roos EM. The impact of physical activity level on the short- and long-term pain relief from supervised exercise therapy and education: a study of 12,796



Danish patients with knee osteoarthritis. *Osteoarthritis and cartilage*. Nov 2018;26(11):1474-1478. doi:10.1016/j.joca.2018.07.010

- 21. Bennell KL, Hunt MA, Wrigley TV, Lim BW, Hinman RS. Role of muscle in the genesis and management of knee osteoarthritis. *Rheumatic diseases clinics of North America*. Aug 2008;34(3):731-54. doi:10.1016/j.rdc.2008.05.005
- 22. Rodriguez-Lopez C, Beckwée D, Luyten FP, Van Assche D, Van Roie E. Reduced knee extensor torque production at low to moderate velocities in postmenopausal women with knee osteoarthritis. *Scand J Med Sci Sports*. Nov 2021;31(11):2144-2155. doi:10.1111/sms.14035
- 23. Skoffer B, Dalgas U, Mechlenburg I, Soballe K, Maribo T. Functional performance is associated with both knee extensor and flexor muscle strength in patients scheduled for total knee arthroplasty: A cross-sectional study. *Journal of rehabilitation medicine*. May 2015;47(5):454-9. doi:10.2340/16501977-1940
- 24. Culvenor AG, Ruhdorfer A, Juhl C, Eckstein F, Øiestad BE. Knee Extensor Strength and Risk of Structural, Symptomatic, and Functional Decline in Knee Osteoarthritis: A Systematic Review and Meta-Analysis. *Arthritis care & research*. May 2017;69(5):649-658. doi:10.1002/acr.23005
- 25. Bryk FF, Dos Reis AC, Fingerhut D, et al. Exercises with partial vascular occlusion in patients with knee osteoarthritis: a randomized clinical trial. *Knee surgery, sports traumatology, arthroscopy*. May 2016;24(5):1580-6. doi:10.1007/s00167-016-4064-7
- 26. Ferraz RB, Gualano B, Rodrigues R, et al. Benefits of Resistance Training with Blood Flow Restriction in Knee Osteoarthritis. *Medicine and science in sports and exercise*. May 2018;50(5):897-905. doi:10.1249/mss.0000000000001530
- 27. Jan MH, Lin JJ, Liau JJ, Lin YF, Lin DH. Investigation of clinical effects of high- and low-resistance training for patients with knee osteoarthritis: a randomized controlled trial. *Physical therapy*. Apr 2008;88(4):427-36. doi:10.2522/ptj.20060300
- 28. Manimmanakorn A, Hamlin MJ, Ross JJ, Taylor R, Manimmanakorn N. Effects of low-load resistance training combined with blood flow restriction or hypoxia on muscle function and performance in netball athletes. *Journal of science and medicine in sport*. Jul 2013;16(4):337-42. doi:10.1016/j.jsams.2012.08.009
- 29. Scott BR, Loenneke JP, Slattery KM, Dascombe BJ. Blood flow restricted exercise for athletes: A review of available evidence. *Journal of science and medicine in sport*. May 2016;19(5):360-7. doi:10.1016/j.jsams.2015.04.014



- 30. Dos Santos LP, Santo R, Ramis TR, Portes JKS, Chakr R, Xavier RM. The effects of resistance training with blood flow restriction on muscle strength, muscle hypertrophy and functionality in patients with osteoarthritis and rheumatoid arthritis: A systematic review with meta-analysis. *PloS one*. 2021;16(11):e0259574. doi:10.1371/journal.pone.0259574
- 31. Giles L, Webster KE, McClelland J, Cook JL. Quadriceps strengthening with and without blood flow restriction in the treatment of patellofemoral pain: a double-blind randomised trial. *Br J Sports Med.* Dec 2017;51(23):1688-1694. doi:10.1136/bjsports-2016-096329
- 32. Grønfeldt BM, Lindberg Nielsen J, Mieritz RM, Lund H, Aagaard P. Effect of bloodflow restricted vs heavy-load strength training on muscle strength: Systematic review and meta-analysis. *Scand J Med Sci Sports*. May 2020;30(5):837-848. doi:10.1111/sms.13632
- 33. Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. *Br J Sports Med.* Jul 2017;51(13):1003-1011. doi:10.1136/bjsports-2016-097071
- 34. Hughes L, Patterson SD. The effect of blood flow restriction exercise on exercise-induced hypoalgesia and endogenous opioid and endocannabinoid mechanisms of pain modulation. *Journal of applied physiology (Bethesda, Md : 1985)*. Apr 1 2020;128(4):914-924. doi:10.1152/japplphysiol.00768.2019
- 35. Lixandrão ME, Ugrinowitsch C, Berton R, et al. Magnitude of Muscle Strength and Mass Adaptations Between High-Load Resistance Training Versus Low-Load Resistance Training Associated with Blood-Flow Restriction: A Systematic Review and Meta-Analysis. *Sports medicine (Auckland, NZ)*. Feb 2018;48(2):361-378. doi:10.1007/s40279-017-0795-y
- 36. Rodrigues R, Ferraz RB, Kurimori CO, et al. Low-Load Resistance Training With Blood-Flow Restriction in Relation to Muscle Function, Mass, and Functionality in Women With Rheumatoid Arthritis. *Arthritis care & research*. Jun 2020;72(6):787-797. doi:10.1002/acr.23911
- 37. Takada S, Okita K, Suga T, et al. Low-intensity exercise can increase muscle mass and strength proportionally to enhanced metabolic stress under ischemic conditions. *Journal of applied physiology (Bethesda, Md : 1985)*. Jul 2012;113(2):199-205. doi:10.1152/japplphysiol.00149.2012
- 38. Yasuda T, Fukumura K, Fukuda T, et al. Muscle size and arterial stiffness after blood flow-restricted low-intensity resistance training in older adults. *Scand J Med Sci Sports*. Oct 2014;24(5):799-806. doi:10.1111/sms.12087



- 39. Centner C, Wiegel P, Gollhofer A, König D. Effects of Blood Flow Restriction Training on Muscular Strength and Hypertrophy in Older Individuals: A Systematic Review and Meta-Analysis. *Sports medicine (Auckland, NZ)*. Jan 2019;49(1):95-108. doi:10.1007/s40279-018-0994-1
- 40. Nielsen JL, Aagaard P, Bech RD, et al. Proliferation of myogenic stem cells in human skeletal muscle in response to low-load resistance training with blood flow restriction. *The Journal of physiology*. Sep 1 2012;590(17):4351-61. doi:10.1113/jphysiol.2012.237008
- 41. Ramos-Campo DJ, Scott BR, Alcaraz PE, Rubio-Arias JA. The efficacy of resistance training in hypoxia to enhance strength and muscle growth: A systematic review and meta-analysis. *European journal of sport science*. Feb 2018;18(1):92-103. doi:10.1080/17461391.2017.1388850
- 42. Jakobsgaard JE, Christiansen M, Sieljacks P, et al. Impact of blood flow-restricted bodyweight exercise on skeletal muscle adaptations. *Clinical physiology and functional imaging*. Feb 15 2018;doi:10.1111/cpf.12509
- 43. Kubo K, Komuro T, Ishiguro N, et al. Effects of low-load resistance training with vascular occlusion on the mechanical properties of muscle and tendon. *J Appl Biomech*. May 2006;22(2):112-9.
- 44. Clarkson MJ, May AK, Warmington SA. Is there rationale for the cuff pressures prescribed for blood flow restriction exercise? A systematic review. *Scand J Med Sci Sports*. Aug 2020;30(8):1318-1336. doi:10.1111/sms.13676
- 45. Næss T. Determining the optimal blood flow restriction protocol for maximising muscle hypertrophy and strength, pressure and cuff width: A mini-review. *J Hum Sport Exerc*. 01/01 2020;16doi:10.14198/jhse.2021.164.02
- 46. Patterson SD, Hughes L, Head P, Warmington S, Brandner C. Blood flow restriction training: a novel approach to augment clinical rehabilitation: how to do it. *Br J Sports Med*. Dec 2017;51(23):1648-1649. doi:10.1136/bjsports-2017-097738
- 47. Patterson SD, Hughes L, Warmington S, et al. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Review. *Front Physiol.* 2019-May-15 2019;10(533)doi:10.3389/fphys.2019.00533
- 48. Vanwye WR, Weatherholt AM, Mikesky AE. Blood Flow Restriction Training: Implementation into Clinical Practice. *Int J Exerc Sci.* 2017;10(5):649-654.
- 49. Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form,



Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). *Arthritis care & research*. Nov 2011;63 Suppl 11:S208-28. doi:10.1002/acr.20632

- 50. Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. *Health and quality of life outcomes*. Nov 3 2003;1:64. doi:10.1186/1477-7525-1-64
- 51. Dobson F, Hinman RS, Roos EM, et al. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis.

  Osteoarthritis and cartilage. Aug 2013;21(8):1042-52. doi:10.1016/j.joca.2013.05.002
- 52. Wright AA, Cook CE, Baxter GD, Dockerty JD, Abbott JH. A comparison of 3 methodological approaches to defining major clinically important improvement of 4 performance measures in patients with hip osteoarthritis. *The Journal of orthopaedic and sports physical therapy*. May 2011;41(5):319-27. doi:10.2519/jospt.2011.3515
- 53. Gill S, McBurney H. Reliability of performance-based measures in people awaiting joint replacement surgery of the hip or knee. *Physiother Res Int*. Sep 2008;13(3):141-52. doi:10.1002/pri.411
- 54. Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. *Research quarterly for exercise and sport*. Jun 1999;70(2):113-9. doi:10.1080/02701367.1999.10608028
- 55. Bennell K, Dobson F, Hinman R. Measures of physical performance assessments: Self-Paced Walk Test (SPWT), Stair Climb Test (SCT), Six-Minute Walk Test (6MWT), Chair Stand Test (CST), Timed Up & Go (TUG), Sock Test, Lift and Carry Test (LCT), and Car Task. *Arthritis care & research*. Nov 2011;63 Suppl 11:S350-70. doi:10.1002/acr.20538
- 56. Coleman G, Dobson F, Hinman RS, Bennell K, White DK. Measures of Physical Performance. *Arthritis care & research*. Oct 2020;72 Suppl 10:452-485. doi:10.1002/acr.24373
- 57. Davey R, Edwards S, Cochrane T. Test–retest Reliability of Lower Extremity Functional and Self-reported Measures in Elderly with Osteoarthritis. *Advances in Physiotherapy*. 12/01 2003;5:155-160. doi:10.1080/1403819038190310017075



- 58. Kennedy DM, Stratford PW, Wessel J, Gollish JD, Penney D. Assessing stability and change of four performance measures: a longitudinal study evaluating outcome following total hip and knee arthroplasty. *BMC musculoskeletal disorders*. 2005/01/28 2005;6(1):3. doi:10.1186/1471-2474-6-3
- 59. Hinarejos P, Goicoechea N, Gidi M, et al. Pressure algometry is a suitable tool to assess anterior knee pain in osteoarthritic patients. *European Journal of Orthopaedic Surgery & Traumatology*. 07/01 2019;29doi:10.1007/s00590-019-02391-w
- 60. Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. Journal of strength and conditioning research. Jan 2009;23(1):312-4. doi:10.1519/jsc.0b013e31818f051c
- 61. Mutlu E, Ozdincler A. Reliability and responsiveness of algometry for measuring pressure pain threshold in patients with knee osteoarthritis. *Journal of physical therapy science*. 06/01 2015;27:1961-5. doi:10.1589/jpts.27.1961
- 62. Pelfort X, Torres-Claramunt R, Sánchez-Soler JF, et al. Pressure algometry is a useful tool to quantify pain in the medial part of the knee: an intra- and inter-reliability study in healthy subjects. *Orthopaedics & traumatology, surgery & research : OTSR*. Sep 2015;101(5):559-63. doi:10.1016/j.otsr.2015.03.016
- 63. Stausholm MB, Bjordal JM, Moe-Nilssen R, Naterstad IF. Pain pressure threshold algometry in knee osteoarthritis: intra- and inter-rater reliability. *Physiotherapy theory and practice*. Jan 12 2022:1-8. doi:10.1080/09593985.2021.2023929
- 64. Wylde V, Palmer S, Learmonth ID, Dieppe P. Test-retest reliability of Quantitative Sensory Testing in knee osteoarthritis and healthy participants. *Osteoarthritis and cartilage*. Jun 2011;19(6):655-8. doi:10.1016/j.joca.2011.02.009
- 65. Beard DJ, Harris K, Dawson J, et al. Meaningful changes for the Oxford hip and knee scores after joint replacement surgery. *J Clin Epidemiol*. Jan 2015;68(1):73-9. doi:10.1016/j.jclinepi.2014.08.009
- 66. Suetta C, Aagaard P, Rosted A, et al. Training-induced changes in muscle CSA, muscle strength, EMG, and rate of force development in elderly subjects after long-term unilateral disuse. *Journal of applied physiology (Bethesda, Md : 1985)*. Nov 2004;97(5):1954-61. doi:10.1152/japplphysiol.01307.2003
- 67. Aagaard P, Andersen JL, Dyhre-Poulsen P, et al. A mechanism for increased contractile strength of human pennate muscle in response to strength training: changes in



muscle architecture. *The Journal of physiology*. Jul 15 2001;534(Pt. 2):613-23. doi:10.1111/j.1469-7793.2001.t01-1-00613.x

- 68. Aagaard P, Simonsen EB, Andersen JL, Magnusson P, Dyhre-Poulsen P. Increased rate of force development and neural drive of human skeletal muscle following resistance training. *Journal of applied physiology (Bethesda, Md : 1985)*. Oct 2002;93(4):1318-26. doi:10.1152/japplphysiol.00283.2002
- 69. Caserotti P, Aagaard P, Larsen JB, Puggaard L. Explosive heavy-resistance training in old and very old adults: changes in rapid muscle force, strength and power. *Scand J Med Sci Sports*. Dec 2008;18(6):773-82. doi:10.1111/j.1600-0838.2007.00732.x
- 70. Bassey EJ, Fiatarone MA, O'Neill EF, Kelly M, Evans WJ, Lipsitz LA. Leg extensor power and functional performance in very old men and women. *Clin Sci (Lond)*. Mar 1992;82(3):321-7. doi:10.1042/cs0820321
- 71. Bassey EJ, Short AH. A new method for measuring power output in a single leg extension: feasibility, reliability and validity. *Eur J Appl Physiol Occup Physiol*. 1990;60(5):385-90. doi:10.1007/bf00713504
- 72. Ahtiainen JP, Hoffren M, Hulmi JJ, et al. Panoramic ultrasonography is a valid method to measure changes in skeletal muscle cross-sectional area. *Eur J Appl Physiol*. Jan 2010;108(2):273-9. doi:10.1007/s00421-009-1211-6
- 73. Mendis MD, Wilson SJ, Stanton W, Hides JA. Validity of real-time ultrasound imaging to measure anterior hip muscle size: a comparison with magnetic resonance imaging. *The Journal of orthopaedic and sports physical therapy*. Sep 2010;40(9):577-81. doi:10.2519/jospt.2010.3286
- 74. Noorkoiv M, Nosaka K, Blazevich AJ. Assessment of quadriceps muscle cross-sectional area by ultrasound extended-field-of-view imaging. *Eur J Appl Physiol*. Jul 2010;109(4):631-9. doi:10.1007/s00421-010-1402-1
- 75. Pinto SS, Cadore EL, Alberton CL, et al. Effects of Intra-session Exercise Sequence during Water-based Concurrent Training. *International journal of sports medicine*. 2014;35(1):41-48.
- 76. Ruas C, Pinto R, D Lima C, Costa P, Brown L. Test-Retest Reliability of Muscle Thickness, Echo-Intensity and Cross Sectional Area of Quadriceps and Hamstrings Muscle Groups Using B-mode Ultrasound. *International Journal of Kinesiology and Sports Science*. 03/11 2017;5:35-41. doi:10.7575/aiac.ijkss.v.5n.1p.35



- 77. Scott JM, Martin DS, Ploutz-Snyder R, et al. Reliability and validity of panoramic ultrasound for muscle quantification. *Ultrasound Med Biol*. Sep 2012;38(9):1656-61. doi:10.1016/j.ultrasmedbio.2012.04.018
- 78. Scott JM, Martin DS, Ploutz-Snyder R, et al. Panoramic ultrasound: a novel and valid tool for monitoring change in muscle mass. *J Cachexia Sarcopenia Muscle*. Jun 2017;8(3):475-481. doi:10.1002/jcsm.12172
- 79. Stokes T, Tripp T, Murphy K, et al. Methodological considerations for and validation of the ultrasonographic determination of human skeletal muscle hypertrophy and atrophy. *Physiological Reports*. 01/01 2021;9doi:10.14814/phy2.14683
- 80. Bergstrom J. MUSCLE ELECTROLYTES IN MAN DETERMINED BY NEUTRON ACTIVATION ANALYSIS ON NEEDLE BIOPSY SPECIMENS. *Scandinavian Journal of Clinical and Laboratory Investigation (England)*. 1962;Vol: 14: Suppl. 68:Medium: X; Size: Pages: 110 2016-06-30.
- 81. Ekblom B. The muscle biopsy technique. Historical and methodological considerations. *Scand J Med Sci Sports*. May 2017;27(5):458-461. doi:10.1111/sms.12808
- 82. Mertz KH, Reitelseder S, Jensen M, et al. Influence of between-limb asymmetry in muscle mass, strength, and power on functional capacity in healthy older adults. *Scand J Med Sci Sports*. Dec 2019;29(12):1901-1908. doi:10.1111/sms.13524
- 83. Nielsen JL, Frandsen U, Jensen KY, et al. Skeletal Muscle Microvascular Changes in Response to Short-Term Blood Flow Restricted Training-Exercise-Induced Adaptations and Signs of Perivascular Stress. *Frontiers in physiology*. 2020;11:556. doi:10.3389/fphys.2020.00556
- 84. Suetta C, Andersen JL, Dalgas U, et al. Resistance training induces qualitative changes in muscle morphology, muscle architecture, and muscle function in elderly postoperative patients. *Journal of applied physiology (Bethesda, Md : 1985)*. Jul 2008;105(1):180-6. doi:10.1152/japplphysiol.01354.2007
- 85. Altman R, Asch E, Bloch D, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. *Arthritis and rheumatism*. Aug 1986;29(8):1039-49. doi:10.1002/art.1780290816
- 86. Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. *Clinical orthopaedics and related research*. Aug 2016;474(8):1886-93. doi:10.1007/s11999-016-4732-4

